CLINICAL TRIAL: NCT05056779
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of Nemolizumab in Subjects With Moderate-to-Severe Atopic Dermatitis With Inadequate Response to or for Whom Cyclosporine A is Not Medically Advisable
Brief Title: Efficacy and Safety of Nemolizumab in Subjects With Moderate-to-Severe Atopic Dermatitis With Inadequate Response to or for Whom Cyclosporine A is Not Medically Advisable
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The study data will not be utilized in the IND and is only being conducted in EU.
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RD.06.SPR.201591; 2021-002166-40 (EudraCT Number)
Record Dates: First submitted 2021-09-15; First posted 2021-09-27 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2021-09

CONDITIONS: Moderate-to-severe Atopic Dermatitis
MeSH Terms: interventions — nemolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nemolizumab (Experimental)
  Interventions: Drug: Nemolizumab
- Placebo (Experimental)
  Interventions: Drug: CD14152 placebo

INTERVENTIONS:
Drug: Nemolizumab — Participants will receive loading dose of 60 milligram (2×30 mg) subcutaneous (SC) injection of nemolizumab at baseline. Thereafter 30 mg nemolizumab will be administered via single SC injection once in 4 week (Q4W) up to week 12.
  Other Names: CD14152
  Arms: Nemolizumab
Drug: CD14152 placebo — Participants will receive loading dose of 60 mg (2×30 mg) SC injection of placebo at baseline. Thereafter 30 mg placebo will be administered via single SC injection Q4W up to week 12.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to investigate the efficacy of nemolizumab administered in combination with topical background therapy (topical corticosteroids [TCS] with or without topical calcineurin inhibitors [TCI]) in adult participants with moderate-to-severe atopic dermatitis (AD) who are not adequately controlled with or are not advised to use oral cyclosporine A (CsA) for medical reasons. The secondary objective is to investigate the safety of nemolizumab in adult participants with moderate-to-severe AD who are not adequately controlled with or are not advised to use oral CsA for medical reasons.

The study will be carried out in up to 70 different locations across Europe.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic AD for at least 2 years before the screening visit and confirmed according to American Academy of Dermatology Consensus at the time of the screening visit.
2. EASI score ≥ 20 at both the screening and baseline visits. Participant with an EASI score of 18-19 at the screening visit only may be reevaluated once within 48 hours.
3. IGA score ≥ 3 (based on the IGA scale ranging from 0 to 4, in which 3 is moderate and 4 is severe) at both the screening and baseline visits.
4. AD involvement ≥ 10% of BSA at both the screening and baseline visits.
5. Documented history by a physician (within 6 months before the screening visit) of inadequate response to topical medications or use of systemic therapies for control of the disease.
6. Agree to apply a moisturizer throughout the study from the screening visit; agree to apply an authorized TCS, with or without TCI, from the screening visit and throughout the study as determined appropriate by the investigator.
7. Documented history of one of the following, where CsA treatment should not be continued/restarted or participant is not currently a candidate for CsA treatment:

   1. Inadequate response to CsA with previous exposure (defined as flare of AD during CsA tapering from a maximum of 6 weeks of high dose [5 mg/kg/day] to maintenance dose [2 to 3 mg/kg/day] or a flare after a minimum of 3 months on maintenance dose). Flare is defined as increase in signs and/or symptoms leading to escalation of therapy (ie, increase in dose, switch to a higher-potency topical corticosteroids [TCS] or start of another systemic nonsteroidal immunosuppressive drug), or
   2. Previous requirement for CsA at doses > 5 mg/kg/day, or duration beyond those specified in the prescribing information (> 1 year)
   3. Intolerance and/or unacceptable toxicity (eg, elevated creatinine, elevated liver function tests, uncontrolled hypertension, paresthesia, headache, nausea, hypertrichosis) with previous CsA exposure
   4. CsA is medically inadvisable due to medical contraindication, use of prohibited medications, risk of AEs (eg, serious infection) or toxicity (eg, renal or liver damage), or hypersensitivity to CsA or excipients, in the opinion of the investigator

   Acceptable documentation includes patient records with information on CsA prescription and treatment outcome, other prohibitive medications/medical history, or written documentation of the conversation with the participant's treating physician, if different than the investigator, as applicable.
8. Other protocol defined inclusion criteria could apply.

Exclusion Criteria:

1. Body weight < 30 kg.
2. One or more of the following criteria at screening or baseline:

   1. Exacerbation of asthma requiring hospitalization in the preceding 12 months.
   2. Asthma that has not been well controlled (i.e, symptoms occurring on > 2 days per week, nighttime awakenings 2 or more times per week, or some interference with normal activities) during the preceding 3 months.
   3. Asthma Control Test (ACT) ≤ 19 (only for subjects with a history of asthma).
   4. Peak expiratory flow (PEF) < 80% of the predicted value.
3. Current medical history of chronic obstructive pulmonary disease and/or chronic bronchitis.
4. Positive serology results (hepatitis B surface antigen [HBsAg] or hepatitis B core antibody [HBcAb], hepatitis C [HCV] antibody with positive HCV RNA, or human immunodeficiency virus [HIV] antibody) at the screening visit.
5. Presence of confounding skin conditions that may interfere with study assessments.
6. Planned or expected major surgical procedure during the clinical study.
7. Other protocol defined exclusion criteria could apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants with Eczema Area and Severity Index-75 (EASI-75) (≥ 75% Improvement in EASI from Baseline) at Week 16 | Week 16
  EASI assesses severity and extent of AD signs through a composite score of erythema, induration/population, excoriation, and lichenification. The severity will be assessed on a scale of 0 (absent) to 3 (severe) for each of the 4 body areas: head/neck, trunk, upper limbs, and lower limbs, with half points allowed. The EASI score can range from 0 to 72 with higher scores representing greater severity of atopic dermatitis.
Proportion of Participants with an Improvement of Peak Pruritus Numeric Rating Scale (PP NRS) ≥ 4 at Week 16 | Week 16
  Pruritus NRS is a scale that will be used by the participants to report the intensity of their pruritus (itch) during the last 24 hours. For maximum itch intensity: the scores are provided on a scale of 0 to 10, with 0 being 'no itch' and 10 being 'worst itch imaginable'. Higher scores indicate worse outcome.

SECONDARY OUTCOMES:
Percent Change from Baseline in EASI at Each Visit Through Week 16 | Baseline through week 16
  EASI assesses severity and extent of AD signs through a composite score of erythema, induration/population, excoriation, and lichenification. The severity will be assessed on a scale of 0 (absent) to 3 (severe) for each of the 4 body areas: head/neck, trunk, upper limbs, and lower limbs, with half points allowed. The EASI score can range from 0 to 72 with higher scores representing greater severity of atopic dermatitis.
Proportion of Participants with at Least 50%, 75%, or 90% Improvement from Baseline in Eczema Area and Severity Index (EASI-50, EASI-75, and EASI-90) at Each Visit Through Week 16 | Baseline through week 16
  EASI assesses severity and extent of AD signs through a composite score of erythema, induration/population, excoriation, and lichenification. The severity will be assessed on a scale of 0 (absent) to 3 (severe) for each of the 4 body areas: head/neck, trunk, upper limbs, and lower limbs, with half points allowed. The EASI score can range from 0 to 72 with higher scores representing greater severity of atopic dermatitis. EASI-50, EASI-75 and EASI-90 responders will be the participants who achieved >=50%, >=75% and >=90% overall improvement in EASI score respectively from baseline to Week 16.
Percent Change From Baseline in Peak Pruritus Numeric Rating Scale (PP NRS) at Each Visit Through Week 16 | Baseline through week 16
  Pruritus NRS is a scale that will be used by the participants to report the intensity of their pruritus (itch) during the last 24 hours. For maximum itch intensity: the scores are provided on a scale of 0 to 10, with 0 being 'no itch' and 10 being 'worst itch imaginable'. Higher scores indicate worse outcome.
Proportion of Participants with an Improvement of Peak Pruritus Numeric Rating Scale (PP NRS) ≥ 4 at Week 1, Week 2, and Each Visit Through Week 16 | From Week 1 to Week 16
  Pruritus NRS is a scale that will be used by the participants to report the intensity of their pruritus (itch) during the last 24 hours. For maximum itch intensity: the scores are provided on a scale of 0 to 10, with 0 being 'no itch' and 10 being 'worst itch imaginable'. Higher scores indicate worse outcome.
Proportion of Participants with Peak Pruritus Numeric Rating Scale (PP NRS) < 2 at each Visit Through Week 16 | Baseline through week 16
  Pruritus NRS is a scale that will be used by the participants to report the intensity of their pruritus (itch) during the last 24 hours. For maximum itch intensity: the scores are provided on a scale of 0 to 10, with 0 being 'no itch' and 10 being 'worst itch imaginable'. Higher scores indicate worse outcome.
Proportion of Participants with an Investigator's Global Assessment (IGA) Success (Defined as an IGA of 0 [Clear] or 1 [Almost clear] and a ≥ 2-Point Reduction from Baseline) at Each Visit Through Week 16 | Baseline through week 16
  IGA is a 5-point scale ranging from 0 (clear) to 4 (severe) used to evaluate the global severity of AD. Higher scores indicate worse outcome.
Proportion of Participants with EASI-75 and improvement of PP NRS ≥ 4 at Each Visit Through Week 16 | Baseline through week 16
  EASI assesses severity and extent of AD signs through a composite score of erythema, induration/population, excoriation, and lichenification. The severity will be assessed on a scale of 0 (absent) to 3 (severe) for each of the 4 body areas: head/neck, trunk, upper limbs, and lower limbs, with half points allowed. The EASI score can range from 0 to 72 with higher scores representing greater severity of atopic dermatitis.
Proportion of Participants with IGA Success and Improvement of PP NRS ≥ 4 at each Visit Through Week 16 | Baseline through week 16
  IGA is a 5-point scale ranging from 0 (clear) to 4 (severe) used to evaluate the global severity of AD. Higher scores indicate worse outcome. Pruritus NRS is a scale that will be used by the participants to report the intensity of their pruritus (itch) during the last 24 hours. For maximum itch intensity: the scores are provided on a scale of 0 to 10, with 0 being 'no itch' and 10 being 'worst itch imaginable'. Higher scores indicate worse outcome.
Proportion of Participants with an Improvement of Sleep Disturbance Numeric Rating Scale (SD NRS) ≥ 4 at Each Visit Through Week 16 | Baseline through week 16
  The sleep disturbance NRS is a scale used by the participants to report the degree of their sleep loss related to AD. Participants will be asked the following questions in their local language: how would you rate your sleep last night? On a scale of 0 to 10, with 0 being 'no sleep loss related to signs/symptoms of AD' and 10 being 'I cannot sleep at all due to the signs/symptoms of AD'. Higher scores indicate worse outcome.
Percent Change from Baseline in Sleep Disturbance Numeric Rating Scale (SD NRS) at Each Visit Through Week 16 | Baseline through week 16
  The sleep disturbance NRS is a scale used by the participants to report the degree of their sleep loss related to AD. Participants will be asked the following questions in their local language: how would you rate your sleep last night? On a scale of 0 to 10, with 0 being 'no sleep loss related to signs/symptoms of AD' and 10 being 'I cannot sleep at all due to the signs/symptoms of AD'. Higher scores indicate worse outcome.
Percent Change from Baseline in SCORing Atopic Dermatitis (SCORAD) and It's Components at Each Visit Through Week 16 | Baseline through week 16
  SCORAD is a clinical tool for assessing the severity and the extent of AD signs and symptoms. Extent and intensity of eczema as well as subjective signs (insomnia, etc.) are assessed and scored. Total score ranges from 0 (absent disease) to 103 (severe disease).
Change from Baseline in Percent of Body Surface Area (BSA) Affected by Atopic Dermatitis (AD) at Each Visit Through Week 16 | Baseline through week 16
Proportion of Participants with Prior Cyclosporine A (CsA) Use Achieving EASI-75 at Each Visit Through Week 16 | Baseline through week 16
  EASI assesses severity and extent of AD signs through a composite score of erythema, induration/population, excoriation, and lichenification. The severity will be assessed on a scale of 0 (absent) to 3 (severe) for each of the 4 body areas: head/neck, trunk, upper limbs, and lower limbs, with half points allowed. The EASI score can range from 0 to 72 with higher scores representing greater severity of atopic dermatitis.
Change from Baseline in Individual Components of the EASI (Averaged Across Body Regions) at Each Visit Through Week 16 | Baseline through week 16
  EASI assesses severity and extent of AD signs through a composite score of erythema, induration/population, excoriation, and lichenification. The severity will be assessed on a scale of 0 (absent) to 3 (severe) for each of the 4 body areas: head/neck, trunk, upper limbs, and lower limbs, with half points allowed. The EASI score can range from 0 to 72 with higher scores representing greater severity of atopic dermatitis.
Change from Baseline in Atopic Dermatitis (AD)-Associated Pain Frequency Through Week 16 | Baseline through week 16
Change from Baseline in Atopic Dermatitis (AD)-Associated Pain Intensity Through Week 16 | Baseline through week 16
Incidence of Rescue Therapy Use Through Week 16 | Baseline through week 16
Change from Baseline in Percentage of Itch-Free Days (Based on PP NRS = 0/1) Through Week 16 | Baseline through week 16
Change from Baseline in Dermatology Life Quality Index (DLQI) Total Score at Each Visit Through Week 16 | Baseline through week 16
  The DLQI is a validated 10-item questionnaire covering domains including symptoms/feelings, daily activities, leisure, work/school, personal relationships, and treatment. The participant will rate each question ranging from 0 (not at all) to 3 (very much) and score ranges from 0 to 30. A higher total score indicates a poorer quality of life (QoL).
Change from Baseline in Patient-Oriented Eczema Measure (POEM) Total Score at Each Visit Through Week 16 | Baseline through week 16
  The POEM is a 7-item questionnaire that assessed disease symptoms (dryness, itching, flaking, cracking, sleep loss, bleeding and weeping) with a scoring system of 0 (absent disease) to 28 (severe disease) (high score indicative of poor quality of life [QOL]).
Number of Days Free of Topical Atopic Dermatitis (AD) Therapy From Baseline to Week 16 | Baseline to Week 16
Change from baseline in Hospital Anxiety and Depression Scale (HADS) for each subscale (ie, depression and anxiety) at each visit through Week 16 | Baseline through week 16
  Hospital Anxiety and Depression Scale (HADS) is a 14-question validated questionnaire completed by the participant for each subscale (i.e. depression and anxiety). Each question has a multiple choice answer which is scored between 0 and 3. Questions are identified as relating to anxiety (A) or depression (D) and a summation for each area is performed leading to a total score of 0 to 21 for each area. Scores of 0 to 7 are considered normal, 8 to 10 are borderline, and >= 11 indicates clinical effects.
Proportion of Participants Reporting Hospital Anxiety and Depression Scale (HADS) anxiety Scores < 8 for those Reporting Scores ≥ 8 at Baseline at Each Visit Through Week 16 | Baseline through week 16
  Hospital Anxiety and Depression Scale (HADS) is a 14-question validated questionnaire completed by the participant for each subscale (i.e. depression and anxiety). Each question has a multiple choice answer which is scored between 0 and 3. Questions are identified as relating to anxiety (A) or depression (D) and a summation for each area is performed leading to a total score of 0 to 21 for each area. Scores of 0 to 7 are considered normal, 8 to 10 are borderline, and >= 11 indicates clinical effects.
Proportion of Participants Reporting HADS depression Scores < 8 for Those Reporting Scores ≥ 8 at Baseline at Each Visit Through Week 16 | Baseline through week 16
  Hospital Anxiety and Depression Scale (HADS) is a 14-question validated questionnaire completed by the participant for each subscale (i.e. depression and anxiety). Each question has a multiple choice answer which is scored between 0 and 3. Questions are identified as relating to anxiety (A) or depression (D) and a summation for each area is performed leading to a total score of 0 to 21 for each area. Scores of 0 to 7 are considered normal, 8 to 10 are borderline, and >= 11 indicates clinical effects.
Change from Baseline in EuroQoL 5-Dimension (EQ-5D) at each visit through Week 16 | Baseline through week 16
  The EQ-5D instrument is a validated questionnaire, completed by the participant that consists of 2 parts. The first part consists of 5 multiple choice QoL questions and the second is a 100 point visual analogue scale (VAS) with 0 being "Worst imaginable health state" and 100 being "Best imaginable health state".
Incidence and Severity of Adverse Events (AEs), Including Adverse Events of Special Interest (AESIs), Treatment Emergent AEs (TEAEs), and serious AEs (SAEs) | Baseline through week 24